CLINICAL TRIAL: NCT05168748
Title: Phase I, Open Label, Multicenter, Dose Escalation and Expansion Study of IMJ995 in Acute Lymphoblastic Leukemia
Brief Title: CD19- and CD22-directed CAR-T Cell Therapy in Patients With Acute Lymphoblastic Leukemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIMJ995A12101; 2021-000677-89 (EudraCT Number)
Record Dates: First submitted 2021-11-03; First posted 2021-12-23 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-09

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: CAR-T; IMJ995; CD19; CD22; acute lymphoblastic leukemia (ALL); pediatric; adolescent
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IMJ995 in ALL (Experimental): Dose escalation and expansion of IMJ995 single agent in ALL
  Interventions: Drug: IMJ995 single agent

INTERVENTIONS:
Drug: IMJ995 single agent — Single intravenous administration of IMJ995

SUMMARY:
This is a first-in-human study to evaluate the feasibility, safety and preliminary antitumor efficacy of autologous chimeric antigen receptor (CAR) T cells targeting both CD19 and CD22, manufactured with T-Charge(TM) process. CAR-T cells will be investigated as single agent in pediatric and adult acute lymphoblastic leukemia (ALL).

DETAILED DESCRIPTION:
This is a phase I, open label, multicenter, dose escalation and expansion study of IMJ995. The study will investigate single agent IMJ995 in two independent groups of acute lymphoblastic leukemia (ALL) patients:

* Pediatric, adolescent and young adult (AYA) ALL patients up to 29 years old
* Adult ALL patients (≥30 years old) safety cohort The pediatric and AYA ALL group consists of two parts: a dose escalation part to evaluate feasibility, characterize safety and identify the recommended dose (RD) of IMJ995, and a dose expansion part to further characterize safety, cellular kinetics and assess preliminary antitumor activity. Once the RD of IMJ995 is determined for this group, the corresponding expansion part may commence.

Once the RD of IMJ995 is determined for the pediatric and AYA group, a safety cohort for adult ALL patients ≥30 years old may commence in parallel to the above mentioned expansion part.

ELIGIBILITY:
Inclusion Criteria:

All patients:

* Evidence of CD19 and/or CD22 cell surface expression on B-ALL blasts in bone marrow or peripheral blood by flow cytometry at time of relapse or prior to study entry.

Pediatric, adolescent and young adult ALL patients:

* 1 - 29 years of age at the time of informed consent form (ICF) signature.
* Relapsed or refractory CD19+ and/or CD22+ ALL after 3 or more lines of treatment OR after allogeneic HCT.
* Must have received a CD19-directed CAR-T treatment (with or without blinatumomab), unless prior loss of CD19 cell surface expression occurred or have not been eligible for CD19 directed CAR-T treatment.
* Lansky (age < 16 years), Karnofsky (age 16-25 years) performance status ≥ 60%. ECOG (age >25 years) performance status that is either 0 or 1 at screening.

Adult ALL patients aged ≥30 years:

* ≥30 years of age at the time of informed consent form (ICF) signature.
* Refractory or relapsed CD19+ and/or CD22+ ALL including at least one of the following:

  * After allogeneic HCT
  * After 2 or more lines of treatment, including blinatumomab and/or inotuzumab
  * Primary refractory disease (defined as failure to achieve a CR at the end of at least 1 induction chemotherapy)
  * First relapse occurring within 12 months from first remission
* ECOG performance status that is either 0 or 1 at screening.

Exclusion Criteria:

* Allogeneic HCT within 12 weeks prior to screening.
* Presence of isolated extra-medullary disease, testicular involvement or bulky disease
* Patients with concomitant genetic syndromes associated with bone marrow failure states: such as patients with Fanconi anemia, Kostmann syndrome, Shwachman syndrome.
* Patients with Burkitt's lymphoma/leukemia
* History of active neurological auto immune or inflammatory disorders

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-24 (Estimated); Primary Completion 2026-08-13 (Estimated); Study Completion 2026-08-13 (Estimated)

PRIMARY OUTCOMES:
Incidence and nature of Dose Limiting Toxicities (Dose Escalation part only, in pediatric, adolescent and young adult ALL patients) | 28 days
  Dose recommendation for IMJ995 in pediatric, adolescent and young adult ALL patients
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) (pediatric, adolescent and young adult ALL patients) | 24 months
  Safety and tolerability
Number of patients infused with planned target dose | 24 months
  Manufacture success rate

SECONDARY OUTCOMES:
Incidence and nature of DLTs during the first 28 days after IMJ995 infusion (safety cohort for adult ALL). | 28 days
  Dose recommendation in adult ALL
Cellular kinetics of IMJ995 (maximum drug concentration - Cmax) | 24 months
  CAR transgene levels will be measured by flow cytometry and quantitative polymerase chain reaction (qPCR) in peripheral blood. PK parameters will be determined using non-compartmental methods for IMJ995.
Cellular kinetics of IMJ995 (area under the drug concentration-time curve - AUC) | 24 months
  CAR transgene levels will be measured by flow cytometry and quantitative polymerase chain reaction (qPCR) in peripheral blood. PK parameters will be determined using non-compartmental methods for IMJ995.
Number of participants with anti-CAR19 and/or anti-CAR22 antibodies | 24 months
  Humoral immunogenicity
Change from baseline in interferon (IFN)-gamma levels in peripheral blood mononuclear cells (PBMCs) | 24 months
  Cellular immunogenicity
Antitumor activity assessed by Complete Remission / Complete Remission with Incomplete Hematologic Recovery (CR/ CRi). | 24 months
  Antitumor activity
Antitumor activity assessed by duration of response. | 24 months
  Duration of response
Incidence and severity of AEs and SAEs after IMJ995 infusion (safety cohort for adult ALL). | 24 months
  Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No